CLINICAL TRIAL: NCT02058381
Title: A Phase Ib Dose De-escalation Study of the Combination of Tamoxifen Plus Goserelin Acetate With Alpelisib (BYL719) or Buparlisib (BKM120) in Premenopausal Patients With Hormone Receptor-positive/HER2-negative Locally Advanced or Metastatic Breast Cancer
Brief Title: A Phase Ib Dose De-escalation Study With BYL719 in Premenopausal Patients With Locally Advanced or Metastatic Breast Cancer
Acronym: B-YOND
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719XIC01
Record Dates: First submitted 2014-01-16; First posted 2014-02-10 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2018-12

CONDITIONS: Pre-menopausal Breast Cancer; PI3K Pathway Inhibition
MeSH Terms: interventions — Alpelisib; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (alpelisib) (Experimental): Alpelisib plus Tamoxifen and Goserelin (Group 1)
  Interventions: Drug: alpelisib (BYL719)
- Group 2 (buparlisib) (Experimental): Buparlisib plus Tamoxifen and Goserelin (Group 2)
  Interventions: Drug: buparlisib (BKM120)

INTERVENTIONS:
Drug: alpelisib (BYL719) — BYL 719 350 mg will be administered orally once daily on a continuous dosing schedule starting on day 1 (Group 1 only).
  Arms: Group 1 (alpelisib)
Drug: buparlisib (BKM120) — BKM120 100 mg will be administered orally once daily on a continuous dosing schedule starting on day 1 (Group 2 only)
  Arms: Group 2 (buparlisib)

SUMMARY:
Based on the evidence acquired in the post-menopausal setting with everolimus and on pre-clinical evidences supporting the investigation of PI3K inhibitors, such as alpelisib and buparlisib, in combination with endocrine therapy in hormone receptor-positive MBC, the purpose of this phase Ib trial is to assess the maximum tolerated dose (MTD) and/or the RP2D(s), to characterize the safety and tolerability, to determine the single and multiple dose PK profile and assess the preliminary anti-tumor activity of alpelisib and buparlisib in combination with tamoxifen plus goserelin acetate in premenopausal hormone receptor-positive advanced breast cancer patientsgroup.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically and/or cytologically confirmed diagnosis of breast cancer
* Patient has radiological or objective evidence of inoperable locally advanced or metastatic breast cancer
* Patient has HER2-negative breast cancer (based on most recently analyzed tumor sample)
* Patient has ER positive and/or PgR positive breast cancer by local laboratory testing
* Patient is premenopausal. Premenopausal status is defined as either:

  1. patient had last menstrual period within the last 12 months, OR
  2. if on tamoxifen within the past 3 months, with a plasma estradiol ≥10 pg/mL and FSH ≤40 IU/l or in the premenopausal range, according to local laboratory definition , OR
  3. in case of chemotherapy induced amenorrhea, with a plasma estradiol ≥10 pg/mL) and/or FSH ≤40 IU/l or in the premenopausal range according to local laboratory definition.
* Patient has no previous history of endocrine therapy in the metastatic setting.

Note:

* Patients who received oral endocrine therapy with duration less than 3 weeks or ≤1 injection of LHRH agonist and discontinued for a reason other than suspicious or evidence of disease progression are eligible
* Adjuvant treatment with tamoxifen monotherapy and LHRH analogue monotherapy is allowed. Patients who received tamoxifen plus LH-RH agonist/antagonist in the adjuvant setting are eligible provided they start investigational treatment at least 12 months after the last dose of tamoxifen or LH-RH agonist/antagonist, whichever came later.
* Patients who were already established on bisphosphonate therapy may continue on bisphosphonates.

  * Patient has received ≤1 prior chemotherapy line for MBC
  * For patient who received prior systemic therapy, radiological or objective evidence of recurrence or progression on or after the last systemic therapy is needed
  * Patient must have as per RECIST 1.1:
* measurable disease or
* non-measurable lytic or mixed (lytic + blastic) bone lesions in the absence of measurable disease.

  * Patient has adequate bone marrow and organ function as defined by the following laboratory values:
  * Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≦ 2 which the investigator believes is stable at the time of screening.
  * Patient has negative serum pregnancy test (β-hCG) within 72 hrs before starting study treatment.

Exclusion criteria

* Patient is post-menopausal.
* Patient has received previous endocrine treatments in the metastatic setting.
* Patient has received previous treatment with PI3K inhibitors, AKT inhibitors, mTOR inhibitors
* Patient has received more than one chemotherapy line for metastatic disease
* Patient has symptomatic CNS metastases
* Patient who has received wide field radiotherapy ≦ 4 weeks or limited field radiation for palliation ≦ 2 weeks prior to starting study drug or who have not recovered to grade 1 or better from related side effects of such therapy (with exception of alopecia alopecia)
* Patient has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
* Patient is currently receiving increasing or chronic treatment (> 5 days) with corticosteroids or another immunosuppressive agent, as chronic administration of corticosteroids (> 5 days) can induce CYP3A4
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
* Patient is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment phase is initiated.
* Patient has a score ≧ 12 on the PHQ-9 questionnaire
* Patient selects a response of "1, 2 or 3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9)
* Patient has a GAD-7 mood scale score ≧ 15
* Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others) or patients with active severe personality disorders (defined according to DSM- IV) are not eligible.
* Patient has ≧ Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety
* Patient has active cardiac disease or a history of cardiac dysfunction
* Patient has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
* Patient has any of the following cardiac conduction abnormalities

  1. Ventricular arrhythmias except for benign premature ventricular contractions
  2. Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  3. Conduction abnormality requiring a pacemaker
  4. Other cardiac arrhythmia not controlled with medication
  5. Patient has a QTcF > 480 msec on the screening ECG (using the QTcF formula)
* Patient is currently receiving treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to treatment start.
* Patient has chronic pulmonary disease including dyspnea at rest from any cause or with interstitial lung disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05-06 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Recommended Phase II Dose (RP2D) | 12 months
  To estimate the MTD(s) and/or the RP2D(s) of a) alpelisib in combination with tamoxifen plus goserelin acetate (Group 1) and b) buparlisib in combination with Tamoxifen plus goserelin acetate (Group 2) in premenopausal hormone receptor-positive locally advanced or MBC patients.

SECONDARY OUTCOMES:
Incidence, type, intensity, severity and seriousness of Adverse Events (AEs) during the first 2 cycles dose interruptions, reductions and dose intensity during the study | 12 months
  To characterize the safety and tolerability of a) alpelisib in combination with tamoxifen plus goserelin acetate and b) buparlisib in combination with Tamoxifen plus goserelin acetate
Alpelisib/buparlisib: plasma concentrations and PK parameters, including but not limited to AUC0-t, AUC0-inf, AUC0-24, Cmax, tmax, CL/F, half-life t1/2 and other PK parameters if deemed appropriate. Tamoxifen: trough plasma concentrations | 12 months
  To determine the single and multiple dose PK profile of a) alpelisib in combination with tamoxifen plus goserelin acetate and b) buparlisib in combination with Tamoxifen plus goserelin acetate
Preliminary anti-tumor activity acccording to RECIST 1.1 : It will include overall response rate, clinical benefit, progression free survival and proportion of patients who are alive without progression at 9 months from the date of treatment start | 12 months
  To assess the preliminary anti-tumor activity of a) alpelisib in combination with tamoxifen plus goserelin acetate and b) buparlisib in combination with Tamoxifen plus goserelin acetate
Index score from the EQ-5D-5L; and WPAI-GH scores for work time missed, impairment while working, overall work impairment, and activity impairment | 12 months
  To evaluate and compare the impact of alpelisib and buparlisib in combination with tamoxifen plus goserelin on patient-reported health status and impact on work using the EQ-5D-5L and WPAI-GH questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Novartis Investigative Site, Hong Kong, Hong Kong
- South Korea (4):
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (5):
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
  - Novartis Investigative Site, New Taipei City, TWN
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

REFERENCES:
- [Derived] Lu YS, Lee KS, Chao TY, Tseng LM, Chitapanarux I, Chen SC, Liu CT, Sohn J, Kim JH, Chang YC, Yang Y, Shotelersuk K, Jung KH, Valenti R, Slader C, Gao M, Park YH. A Phase Ib Study of Alpelisib or Buparlisib Combined with Tamoxifen Plus Goserelin in Premenopausal Women with HR-Positive HER2-Negative Advanced Breast Cancer. Clin Cancer Res. 2021 Jan 15;27(2):408-417. doi: 10.1158/1078-0432.CCR-20-1008. Epub 2020 Jul 27. PMID 32718997